CLINICAL TRIAL: NCT05095012
Title: Implementation of a Clinical Pathway for Paediatric Concussion in Acute Care Settings: Measuring Health Outcomes of the RECOVER Intervention Project
Brief Title: RECOVER Clinical Pathway for Pediatric Concussion
Acronym: RECOVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Brain Canada (Other); Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: REB18-0405
Record Dates: First submitted 2021-09-08; First posted 2021-10-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2021-08

CONDITIONS: Concussion, Brain; Pediatric Disorder; Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: The project will involve a stepped wedge time series design to evaluate the implementation of the Maternal Newborn and Child Health clinical pathway for the acute care of pediatric concussion.
Masking Description: Each site will be randomized to a start date. Once a site starts the clinical pathway, the clinical pathway tools (assessment, education and referral tools) will be utilized by staff in that particular emergency department. Patients and parents will be unaware of clinical pathway.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical Pathway Participation (Other): Patients that are seen in an emergency department participating in the clinical pathway will not be aware of any changes, other than be given a specific education handout at discharge and be advised to visit the recoverconcussion.ca web portal. Specialty referrals for high risk patients will automatically be made during the emergency visit, through the clinical pathway.
  Interventions: Other: Pediatric Acute Care Concussion Clinical Pathway

INTERVENTIONS:
Other: Pediatric Acute Care Concussion Clinical Pathway — MD assessment will be partially standardized to assess for patients at higher risk of becoming persistently symptomatic. These patients scoring as 'high risk' will be referred to one of three specialty clinics. High risk is defined as scoring 9 or higher out of 12 on the 5P score.

SUMMARY:
The project encompasses the development and implementation of an acute care, pediatric concussion clinical pathway at 5 pediatric emergency departments in the province of Alberta (Canada).

DETAILED DESCRIPTION:
Clinical pathways (CPs) do not currently guide the care of children with concussions presenting to acute care settings in Alberta. The Alberta Health Services Maternal Newborn Child & Youth (MNCY) Strategic Clinical Network established a work group to develop best-practice, evidence-based Clinical Practice Guidelines for the management of concussion that are being translated into specific CPs for different clinical settings.

The research has three key objectives:

1. Design an evidence-based, knowledge-user informed, and theory-driven approach to implementation of a clinical pathway for acute care of pediatric concussion. Guided by the Theoretical Domains Framework (TDF), the investigators will assess barriers and facilitators likely to influence uptake of the CP in acute care settings. The results of that assessment will inform implementation strategy design, again guided by the TDF.
2. Evaluate the impact of the implementation of the CP on patient-centered outcomes using a stepped wedge cluster randomised trial. Within the context of a stepped wedge cluster randomised trial, the investigators will assess relevant process and clinical outcomes to determine whether implementation of the CP results in significant uptake of the pathway, as well as higher patient satisfaction and better health outcomes following concussion.
3. Determine whether the implementation and use of a CP for acute care of pediatric concussion is associated with changes in health care utilization and associated costs. Health care utilization and costs associated with care of concussion will be compared before and after the implementation of the CP. Utilization and costs are expected to remain stable or decline following implementation of the CP.

ELIGIBILITY:
Inclusion Criteria:

* Children evaluated for concussion (including their parents) January 30 - November 30, 2019 at the 5 participating emergency departments

Exclusion Criteria:

* moderate to severe brain injury

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2878 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Process Outcome | Through study enrollment (Jan 30 - Nov 30, 2019) 11 months
  Measurement of clinician utilization of the newly implemented clinical pathway. Clinician utilization was represented by proportion of clinician-completed 5P assessments per diagnosed concussion. Data was also collected on the number of high risk referrals made through the clinical pathway and the number of handouts provided by the clinician to patients and families.
Clinical Outcome | Through study enrollment, plus a 6 follow-up period, 15 months
  Time to symptom resolution using weekly ratings by patients and parents of whether patient has returned to pre-injury status. Parents and children were asked asked to complete a numeric scale of 0 to 10 (where 0 is very bad and 10 is back to normal), how do you feel now?

SECONDARY OUTCOMES:
Emergency Department satisfaction | Through study enrollment (Jan 30 - Nov 30, 2019) 11 months
  Ratings of care received in the emergency department
RECOVER web portal usage | 1 year
  Number of unique website hits per IP address
Adherence to discharge recommendations | Through study enrollment (Jan 30 - Nov 30, 2019) 11 months
  Rate of patient and parent reported adherence to physician discharge instructions
Rate of diagnosed concussions | Through study enrollment (Jan 30 - Nov 30, 2019) 11 months
  Rate of diagnosed concussions per visit (as noted by billing codes)
Rate of Head CT scans ordered | Through study enrollment (Jan 30 - Nov 30, 2019) 11 months
  Rate of CT scans ordered per diagnosed concussion
Post-concussive symptom ratings | Through study enrollment (Jan 30 - Nov 30, 2019) 11 months
  Child and parent symptoms ratings measured using the Health and Behaviour Inventory. Measured weekly from injury to resolution of symptoms.
Quality of life ratings | 4 weeks post injury
  Child and parent quality of life ratings measured by the Pediatric Quality of Life Inventory

OTHER OUTCOMES:
Health care utilization 1: Acute care length of stay | Through study enrollment (Jan 30 - Nov 30, 2019) 11 months
  Duration of stay in the emergency department
Health care utilization 2: Return visits within 72 hours of discharge | Within 72 hours of initial discharge from the emergency department
  Numbers of patients that returned back to the emergency department for a subsequent visit
Health care utilization 3: Number of subsequent outpatient visits | Within 3 months of initial discharge from the emergency department
  Number of outpatient medical visits attended by patients
Health care costs | Through study enrollment, plus a 3 follow-up period, 14 months
  Cost of emergency department visit(s) and subsequent outpatient visits as determined by administrative data

CONTACTS AND LOCATIONS:
Overall Officials: Keith Yeates, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ly A, Zemek R, Wright B, Zwicker J, Schneider K, Mikrogianakis A, Conradi A, Johnson D, Clark B, Barlow K, Burey J, Kolstad A, Yeates KO. "What is the actual goal of the pathway?": examining emergency department physician and nurse perspectives on the implementation of a pediatric concussion pathway using the theoretical domains framework. BMC Health Serv Res. 2021 Feb 5;21(1):119. doi: 10.1186/s12913-021-06110-2. PMID 33546684
- [Derived] Yeates KO, Barlow KM, Wright B, Tang K, Barrett O, Berdusco E, Black AM, Clark B, Conradi A, Godfrey H, Kolstad AT, Ly A, Mikrogianakis A, Purser R, Schneider K, Stang AS, Zemek R, Zwicker JD, Johnson DW. Health care impact of implementing a clinical pathway for acute care of pediatric concussion: a stepped wedge, cluster randomised trial. CJEM. 2023 Jul;25(7):627-636. doi: 10.1007/s43678-023-00530-1. Epub 2023 Jun 23. PMID 37351798

DOCUMENTS (2):
  • Study Protocol (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT05095012/Prot_001.pdf
  • Informed Consent Form (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT05095012/ICF_000.pdf